CLINICAL TRIAL: NCT06776341
Title: Retrospective and Longitudinal Prospective Natural History Study of GEMIN5-Related Neurodevelopmental Disorder
Brief Title: Natural History Study of GEMIN-5 Related Neurodevelopmental Disorder
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kate Kielty, Principal Investigator, University of Pittsburgh
Other Study IDs: STUDY24060013
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: SMN Complex Proteins; GEMIN5 Protein, Human; Neurodevelopmental Disorders
Keywords: GEMIN5; Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 26 Years
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GEMIN5: GEMIN5
  Interventions: Other: GEMIN5-Related Neurodevelopmental Disorder

INTERVENTIONS:
Other: GEMIN5-Related Neurodevelopmental Disorder — This is an observational study. The investigators will collect data from participants' medical records regarding neurodevelopmental outcomes (eg. cognitive, speech and language, motor skills, developmental skills, vision, hearing), Time to event (Acquistion and loss of developmental milestones), and, if available, data regarding MRIs (presence of cerebellar atrophy), survival, visiion, hearing, and biomarkers of disease.

SUMMARY:
This study will include a comprehensive retrospective chart review and a longitudinal prospective observational natural history study to characterize the phenotypic spectrum of GEMIN5-Related Neurodevelopmental Disorder. We aim to define the trajectory of this ultra-rare disease, core clinical features, characteristics at disease onset and diagnosis, neurological symptomatology, and neuroimaging findings over time. In this study, biological specimens (serum) will also be collected in a biorepository for translational research purposes.

DETAILED DESCRIPTION:
This study will include individuals across the lifespan with molecularly confirmed GEMIN5 biallelic mutations.

This study will be ongoing indefinitely.

There are three main components to the study as are detailed below:

1. A retrospective chart review of UPMC medical records and other institutions' medical records, for all patients in the study. Families/patients will provide staff with a signed Release of Information, so that we can obtain a copy of the participants complete medical record which will be requested from previously treating physicians. This may include records from several disciplines, for example neurological and physical exams, neurodevelopmental testing (cognitive, motor, language and daily living skills), growth parameters, results to previous genetic testing, MRI, lab results including lumbar puncture studies, audiologic exam, vision screening, nerve conduction studies, ophthalmologic exam, swallow studies, co-morbidities, and family history.
2. An observational, longitudinal prospective study of patients seen at the UPMC Center for Neuogenomics (CCNG) clinic. Clinical data obtained as part of a typical CCNG visit include vital signs, measurements (weight, head circumference, length), a developmental history, neurodevelopmental testing (eg. cognitive, speech and language, motor skills, developmental skills, vision, hearing), and a comprehensive neurological exam, including an ataxia rating scale. Additionally, any neurodiagnostic results obtained clinically are reviewed if available, such as MRI brain and spine, EEG, and nerve conductions studies.
3. Patients who are seen at the CCNG clinic in person may opt to submit an optional research biological samples.

Primary endpoint:

Neurodevelopmental outcomes

Secondary endpoint (if available):

MRI - presence of cerebellar atrophy Survival Vision Hearing Biomarkers of disease

ELIGIBILITY:
Inclusion Criteria:

* Individuals with molecularly confirmed GEMIN5 biallelic mutations, ages 0 years and above

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with GEMIN5-Related Neurodevelopmental Disorder
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
neurodevelopmental outcomes | 26 years
  time to acquisition and/or loss of milestones

SECONDARY OUTCOMES:
MRI | 26 years
  presence of cerebellar atrophy
Survival | 26 years
  age at death
Vision | 26 years
  presence of ocular pathology
Hearing | 26 years
  presence of hearing loss
Biomarkers of disease | 26 years
  Biomarkers of disease

CONTACTS AND LOCATIONS:
Overall Officials: Kate Kielty, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No